CLINICAL TRIAL: NCT02104817
Title: A Long-Term Outcomes Study to Assess STatin Residual Risk Reduction With EpaNova in HiGh Cardiovascular Risk PatienTs With Hypertriglyceridemia (STRENGTH)
Brief Title: Outcomes Study to Assess STatin Residual Risk Reduction With EpaNova in HiGh CV Risk PatienTs With Hypertriglyceridemia
Acronym: STRENGTH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: The Cleveland Clinic (Other); IQVIA RDS Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D5881C00004; 2014-001069-28 (EudraCT Number)
Record Dates: First submitted 2014-04-02; First posted 2014-04-04 (Estimated); Results first posted 2021-07-28 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Eligible Men or Women Considered High Risk for Atherosclerotic Cardiovascular Disease (CVD)
Keywords: omega-3 carboxylic acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EPANOVA (Experimental): Epanova + statin, once daily
  Interventions: Drug: Epanova® (omega-3 carboxylic acids)
- Corn oil (Active Comparator): Corn oil + Statin
  Interventions: Drug: corn oil control

INTERVENTIONS:
Drug: Epanova® (omega-3 carboxylic acids) — Adjunct to statin therapy and diet in high risk adult patients for the prevention and reduction of major adverse cardiovascular events (MACE)
  Other Names: omega-3 carboxylic acids
  Arms: EPANOVA
Drug: corn oil control — corn oil control arm
  Arms: Corn oil

SUMMARY:
The study is a randomized, double-blind, placebo-controlled (corn oil), parallel group design that will enroll approximately 13,000 patients with hypertriglyceridemia and low HDL and high risk for CVD to be randomized 1:1 to either corn oil + statin or Epanova + statin, once daily, for approximately 3-5 years as determined when the number of MACE outcomes is reached.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women, ≥18 years of age.
2. Patient must be on a stable diet and statin* therapy at least 4 weeks prior to randomization (Visit 2) and meet the following criteria:

   1. LDL-C <100 mg/dL
   2. TG level ≥180 and <500 mg/dL and HDL-C <42 mg/dL for men or HDL-C <47 mg/dL for women
3. Patient is at high risk for a future cardiovascular event if at least one of the following criteria (3a, 3b or 3c)* is present via patient history, physical exam, or medical records at the time of screening:

   1. Any atherosclerotic CVD as defined in protocol.
   2. History of diabetes mellitus (type 1 or 2) and ≥40 years of age for men and ≥50 years of age for women, plus one of the risk factors defined in protocol.
   3. Male patients >50 years of age or females >60 years of age, with at least one of the risk factors defined in protocol.

Key Exclusion Criteria:

1. Allergy or intolerance to omega-3 carboxylic acids, omega-3 fatty acids, omega-3-acid ethyl esters, or corn oil. 2.Use of fibrates, bile acid sequestrants, or niacin or its analogues (>250 mg/day) within 4 weeks prior to Visit 2. 3.Statin naïve at Visit 1.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13078 (Actual)
Dates: Start 2014-10-30 (Actual); Primary Completion 2020-05-27 (Actual); Study Completion 2020-05-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Nissen, MD, Principal Investigator — The Cleveland Clinic; Michael Lincoff, MD, Principal Investigator — The Cleveland Clinic; Stephen Nicholls, MD, Principal Investigator — MonashHeart
Locations (509):
- United States (186):
  - Research Site, Birmingham, Alabama
  - Research Site, Huntsville, Alabama
  - Research Site, Muscle Shoals, Alabama
  - Research Site, Chandler, Arizona
  - Research Site, Gilbert, Arizona
  - Research Site, Glendale, Arizona
  - Research Site, Mesa, Arizona
  - Research Site, Phoenix, Arizona
  - Research Site, Tempe, Arizona
  - Research Site, Tucson, Arizona
  - Research Site, Little Rock, Arkansas
  - Research Site, Carlsbad, California
  - Research Site, Fresno, California
  - Research Site, Greenbrae, California
  - Research Site, Long Beach, California
  - Research Site, Los Angeles, California
  - Research Site, Milpitas, California
  - Research Site, Newport Beach, California
  - Research Site, Northridge, California
  - Research Site, Palm Springs, California
  - Research Site, San Diego, California
  - Research Site, Santa Ana, California
  - Research Site, Santa Rosa, California
  - Research Site, Tarzana, California
  - Research Site, Colorado Springs, Colorado
  - Research Site, Denver, Colorado
  - Research Site, Waterbury, Connecticut
  - Research Site, Boca Raton, Florida
  - Research Site, Clearwater, Florida
  - Research Site, Coral Gables, Florida
  - Research Site, Davie, Florida
  - Research Site, Delray Beach, Florida
  - Research Site, Fort Lauderdale, Florida
  - Research Site, Hialeah, Florida
  - Research Site, Homestead, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Lake Worth, Florida
  - Research Site, Lakeland, Florida
  - Research Site, Miami, Florida
  - Research Site, New Port Richey, Florida
  - Research Site, Pembroke Pines, Florida
  - Research Site, Pensacola, Florida
  - Research Site, Pinellas Park, Florida
  - Research Site, Port Charlotte, Florida
  - Research Site, Spring Hill, Florida
  - Research Site, Tamarac, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Marietta, Georgia
  - Research Site, Sandy Springs, Georgia
  - Research Site, Savannah, Georgia
  - Research Site, Arlington Heights, Illinois
  - Research Site, Blue Island, Illinois
  - Research Site, Champaign, Illinois
  - Research Site, Chicago, Illinois
  - Research Site, Evanston, Illinois
  - Research Site, Naperville, Illinois
  - Research Site, Oakbrook Terrace, Illinois
  - Research Site, Sterling, Illinois
  - Research Site, Anderson, Indiana
  - Research Site, Avon, Indiana
  - Research Site, Elkhart, Indiana
  - Research Site, Evansville, Indiana
  - Research Site, Fort Wayne, Indiana
  - Research Site, Franklin, Indiana
  - Research Site, Greenfield, Indiana
  - Research Site, Muncie, Indiana
  - Research Site, Valparaiso, Indiana
  - Research Site, Iowa City, Iowa
  - Research Site, Augusta, Kansas
  - Research Site, Overland Park, Kansas
  - Research Site, Louisville, Kentucky
  - Research Site, Monroe, Louisiana
  - Research Site, Shreveport, Louisiana
  - Research Site, Slidell, Louisiana
  - Research Site, Auburn, Maine
  - Research Site, Baltimore, Maryland
  - Research Site, Elkridge, Maryland
  - Research Site, Hyannis, Massachusetts
  - Research Site, Quincy, Massachusetts
  - Research Site, Bay City, Michigan
  - Research Site, Cadillac, Michigan
  - Research Site, Kalamazoo, Michigan
  - Research Site, Saginaw, Michigan
  - Research Site, Traverse City, Michigan
  - Research Site, Edina, Minnesota
  - Research Site, Minneapolis, Minnesota
  - Research Site, Port Gibson, Mississippi
  - Research Site, Tupelo, Mississippi
  - Research Site, Bridgeton, Missouri
  - Research Site, Hazelwood, Missouri
  - Research Site, Omaha, Nebraska
  - Research Site, Las Vegas, Nevada
  - Research Site, Bridgewater, New Jersey
  - Research Site, Camden, New Jersey
  - Research Site, Elmer, New Jersey
  - Research Site, Haddon Heights, New Jersey
  - Research Site, Sewell, New Jersey
  - Research Site, Sicklerville, New Jersey
  - Research Site, Albany, New York
  - Research Site, Binghamton, New York
  - Research Site, Laurelton, New York
  - Research Site, Lawrence, New York
  - Research Site, New York, New York
  - Research Site, Saratoga Springs, New York
  - Research Site, Southampton, New York
  - Research Site, Troy, New York
  - Research Site, Asheville, North Carolina
  - Research Site, Cary, North Carolina
  - Research Site, Charlotte, North Carolina
  - Research Site, Greensboro, North Carolina
  - Research Site, Greenville, North Carolina
  - Research Site, Hickory, North Carolina
  - Research Site, Mooresville, North Carolina
  - Research Site, Morganton, North Carolina
  - Research Site, Raleigh, North Carolina
  - Research Site, Rocky Mount, North Carolina
  - Research Site, Salisbury, North Carolina
  - Research Site, Wilmington, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Grand Forks, North Dakota
  - Research Site, Akron, Ohio
  - Research Site, Cincinnati, Ohio
  - Research Site, Cleveland, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Marion, Ohio
  - Research Site, Maumee, Ohio
  - Research Site, Middleburg Hts, Ohio
  - Research Site, Midwest City, Oklahoma
  - Research Site, Norman, Oklahoma
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Bend, Oregon
  - Research Site, Corvallis, Oregon
  - Research Site, Portland, Oregon
  - Research Site, Allentown, Pennsylvania
  - Research Site, Beaver, Pennsylvania
  - Research Site, Danville, Pennsylvania
  - Research Site, Doylestown, Pennsylvania
  - Research Site, Ephrata, Pennsylvania
  - Research Site, Flourtown, Pennsylvania
  - Research Site, Johnstown, Pennsylvania
  - Research Site, Natrona Heights, Pennsylvania
  - Research Site, Newport, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Port Matilda, Pennsylvania
  - Research Site, Tipton, Pennsylvania
  - Research Site, Wilkes-Barre, Pennsylvania
  - Research Site, Anderson, South Carolina
  - Research Site, Charleston, South Carolina
  - Research Site, Fountain Inn, South Carolina
  - Research Site, Greer, South Carolina
  - Research Site, Mt. Pleasant, South Carolina
  - Research Site, Rock Hill, South Carolina
  - Research Site, Simpsonville, South Carolina
  - Research Site, Spartanburg, South Carolina
  - Research Site, Rapid City, South Dakota
  - Research Site, Bristol, Tennessee
  - Research Site, Chattanooga, Tennessee
  - Research Site, Johnson City, Tennessee
  - Research Site, Kingsport, Tennessee
  - Research Site, Knoxville, Tennessee
  - Research Site, Arlington, Texas
  - Research Site, Austin, Texas
  - Research Site, Corpus Christi, Texas
  - Research Site, Dallas, Texas
  - Research Site, Fort Worth, Texas
  - Research Site, Houston, Texas
  - Research Site, Irving, Texas
  - Research Site, Mission, Texas
  - Research Site, Odessa, Texas
  - Research Site, Plano, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Victoria, Texas
  - Research Site, Clinton, Utah
  - Research Site, Ogden, Utah
  - Research Site, Orem, Utah
  - Research Site, Salt Lake City, Utah
  - Research Site, Burke, Virginia
  - Research Site, Danville, Virginia
  - Research Site, Herndon, Virginia
  - Research Site, Lynchburg, Virginia
  - Research Site, Manassas, Virginia
  - Research Site, Port Orchard, Washington
  - Research Site, Green Bay, Wisconsin
  - Research Site, La Crosse, Wisconsin
  - Research Site, Madison, Wisconsin
  - Research Site, Wausau, Wisconsin
- Australia (14):
  - Research Site, Adelaide
  - Research Site, Blacktown
  - Research Site, Box Hill
  - Research Site, Cowra
  - Research Site, Forbes
  - Research Site, Fremantle
  - Research Site, Herston
  - Research Site, Joondalup
  - Research Site, Maroubra
  - Research Site, Milton
  - Research Site, South Brisbane
  - Research Site, Southport
  - Research Site, Tumbi Vmbi
  - Research Site, Wollongong
- Belgium (10):
  - Research Site, Aalst
  - Research Site, Antwerp
  - Research Site, Bruges
  - Research Site, Brussels
  - Research Site, Genk
  - Research Site, Halen
  - Research Site, Leuven
  - Research Site, Liège
  - Research Site, Mol
  - Research Site, Mons
- Canada (17):
  - Research Site, New Westminster, British Columbia
  - Research Site, Vancouver, British Columbia
  - Research Site, Barrie, Ontario
  - Research Site, Brampton, Ontario
  - Research Site, Cambridge, Ontario
  - Research Site, Etobicoke, Ontario
  - Research Site, Newmarket, Ontario
  - Research Site, North York, Ontario
  - Research Site, Peterborough, Ontario
  - Research Site, Thornhill, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Granby, Quebec
  - Research Site, Laval, Quebec
  - Research Site, Longueuil, Quebec
  - Research Site, Mirabel, Quebec
  - Research Site, Québec, Quebec
  - Research Site, Sherbrooke, Quebec
- China (27):
  - Research Site, Beijing
  - Research Site, Changchun
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Chongqing
  - Research Site, Guangzhou
  - Research Site, Haerbin
  - Research Site, Haikou
  - Research Site, Hohhot
  - Research Site, Jilin
  - Research Site, Lanzhou
  - Research Site, Nanchang
  - Research Site, Nanjing
  - Research Site, Nanning
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Suzhou
  - Research Site, Taiyuan
  - Research Site, Tianjin
  - Research Site, Ürümqi
  - Research Site, Xi'an
  - Research Site, Xuzhou
  - Research Site, Yanji
  - Research Site, Yinchuan
  - Research Site, Yueyang
  - Research Site, Zhanjiang
  - Research Site, Zhenjiang
- Czechia (18):
  - Research Site, Beroun
  - Research Site, Brno
  - Research Site, Choceň
  - Research Site, Chrudim
  - Research Site, Hodonín
  - Research Site, Hostivice
  - Research Site, Hradec Králové
  - Research Site, Jindřichův Hradec
  - Research Site, Olomouc
  - Research Site, Ostrava
  - Research Site, Pardubice
  - Research Site, Prague
  - Research Site, Praha 10 - Strasnice
  - Research Site, Přerov
  - Research Site, Slaný
  - Research Site, Trutnov
  - Research Site, Třemošná
  - Research Site, Zlín
- Denmark (7):
  - Research Site, Aalborg
  - Research Site, Århus N
  - Research Site, Hellerup
  - Research Site, Herlev
  - Research Site, København Ø
  - Research Site, Svendborg
  - Research Site, Viborg
- Estonia (4):
  - Research Site, Haabneeme
  - Research Site, Pärnu
  - Research Site, Tallinn
  - Research Site, Tartu
- Hungary (26):
  - Research Site, Baja
  - Research Site, Balatonfüred
  - Research Site, Balatongyörök
  - Research Site, Ballasagyarmat
  - Research Site, Békéscsaba
  - Research Site, Budapest
  - Research Site, Csorna
  - Research Site, Debrecen
  - Research Site, Eger
  - Research Site, Gödöllő
  - Research Site, Gyula
  - Research Site, Hajdúszoboszló
  - Research Site, Hatvan
  - Research Site, Kalocsa
  - Research Site, Kiskunhalas
  - Research Site, Komárom
  - Research Site, Létavértes
  - Research Site, Mohács
  - Research Site, Nagykanizsa
  - Research Site, Nyíregyháza
  - Research Site, Szeged
  - Research Site, Szekszárd
  - Research Site, Szentes
  - Research Site, Székesfehérvár
  - Research Site, Veszprém
  - Research Site, Zalaegerszeg
- Italy (14):
  - Research Site, Bergamo
  - Research Site, Bologna
  - Research Site, Brescia
  - Research Site, Cinisello Balsamo
  - Research Site, Cona
  - Research Site, L’Aquila
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Parma
  - Research Site, Pavia
  - Research Site, Perugia
  - Research Site, Roma
  - Research Site, San Giovanni Rotondo
  - Research Site, Trieste
- Japan (43):
  - Research Site, Adachi-ku
  - Research Site, Akishima-shi
  - Research Site, Akita
  - Research Site, Amagasaki-shi
  - Research Site, Chikushi-gun
  - Research Site, Chikushino-shi
  - Research Site, Chūōku
  - Research Site, Fujisawa-shi
  - Research Site, Gifu
  - Research Site, Hachioji-shi
  - Research Site, Hakusan-shi
  - Research Site, Ichikawa-shi
  - Research Site, Imabari
  - Research Site, Itoshima-shi
  - Research Site, Kasugai-shi
  - Research Site, Kawanishi-shi
  - Research Site, Kishiwada-shi
  - Research Site, Kitakyushu-shi
  - Research Site, Kochi
  - Research Site, Kyoto
  - Research Site, Maebashi
  - Research Site, Matsudo-shi
  - Research Site, Matsumoto-shi
  - Research Site, Matsuyama
  - Research Site, Meguro-ku
  - Research Site, Minatoku
  - Research Site, Nagoya
  - Research Site, Nakagami-gun
  - Research Site, Niigata
  - Research Site, Onga-gun
  - Research Site, Osaka
  - Research Site, Ōita
  - Research Site, Saga
  - Research Site, Sapporo
  - Research Site, Sendai
  - Research Site, Shinagawa-ku
  - Research Site, Shinjuku-ku
  - Research Site, Takamatsu
  - Research Site, Takasaki-shi
  - Research Site, Tokorozawa-shi
  - Research Site, Toshima-ku
  - Research Site, Tsuchiura-shi
  - Research Site, Yokohama
- Lithuania (6):
  - Research Site, Alytus
  - Research Site, Kaunas
  - Research Site, Klaipėda
  - Research Site, Panevezys
  - Research Site, Šiauliai
  - Research Site, Vilnius
- Mexico (8):
  - Research Site, Chihuahua City
  - Research Site, Cuautitlán Izcalli
  - Research Site, Culiacán
  - Research Site, Guadalajara
  - Research Site, Mérida
  - Research Site, México
  - Research Site, Monterrey
  - Research Site, Zapopan, Jalisco
- Netherlands (25):
  - Research Site, Almelo
  - Research Site, Almere Stad
  - Research Site, Amsterdam
  - Research Site, Apeldoorn
  - Research Site, Arnhem
  - Research Site, Beek
  - Research Site, Delft
  - Research Site, Ede
  - Research Site, Eindhoven
  - Research Site, Harderwijk
  - Research Site, Heerlen
  - Research Site, Hilversum
  - Research Site, Hoofddorp
  - Research Site, Hoogeveen
  - Research Site, Hoorn
  - Research Site, Maastricht
  - Research Site, Nijmegen
  - Research Site, Rotterdam
  - Research Site, Schiedam
  - Research Site, Sneek
  - Research Site, Tilburg
  - Research Site, Utrecht
  - Research Site, Venlo
  - Research Site, Zoetermeer
  - Research Site, Zwijndrecht
- New Zealand (5):
  - Research Site, Auckland
  - Research Site, Christchurch
  - Research Site, Havelock North
  - Research Site, Rotorua
  - Research Site, Wellington
- Poland (24):
  - Research Site, Bialystok
  - Research Site, Chorzów
  - Research Site, Elblag
  - Research Site, Gdansk
  - Research Site, Gdynia
  - Research Site, Katowice
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Lublin
  - Research Site, Oświęcim
  - Research Site, Parczew
  - Research Site, Piaseczno
  - Research Site, Poznan
  - Research Site, Puławy
  - Research Site, Ruda Śląska
  - Research Site, Rzeszów
  - Research Site, Sobótka
  - Research Site, Sopot
  - Research Site, Staszów
  - Research Site, Torun
  - Research Site, Warsaw
  - Research Site, Wroclaw
  - Research Site, Zamość
  - Research Site, Zgierz
- Russia (12):
  - Research Site, Barnaul
  - Research Site, Kemerovo
  - Research Site, Moscow
  - Research Site, Novosibirsk
  - Research Site, Omsk
  - Research Site, Orenburg
  - Research Site, Perm
  - Research Site, Rostov-on-Don
  - Research Site, Ryazan
  - Research Site, Saint Petersburg
  - Research Site, Tomsk
  - Research Site, Yaroslavl
- South Africa (22):
  - Research Site, Bloemfontein
  - Research Site, Breyten
  - Research Site, Brits
  - Research Site, Cape Town
  - Research Site, Centurion
  - Research Site, Durban
  - Research Site, George
  - Research Site, Johannesburg
  - Research Site, Krugersdorp
  - Research Site, Kuilsrivier
  - Research Site, KwaDukuza
  - Research Site, Mamelodi East
  - Research Site, Middelburg
  - Research Site, Moloto South
  - Research Site, Paarl
  - Research Site, Port Elizabeth
  - Research Site, Potchefstroom
  - Research Site, Pretoria
  - Research Site, Somerset West
  - Research Site, Soweto
  - Research Site, Verulam
  - Research Site, Worcester
- South Korea (6):
  - Research Site, Busan
  - Research Site, Gwangju
  - Research Site, Incheon
  - Research Site, Seongnam-si
  - Research Site, Seoul
  - Research Site, Ulsan
- Taiwan (2):
  - Research Site, Kaohsiung City
  - Research Site, Taipei
- Ukraine (13):
  - Research Site, Cherkasy
  - Research Site, Ivano-Frankivsk
  - Research Site, Kharkiv Region
  - Research Site, Kyiv
  - Research Site, Lutsk
  - Research Site, Lviv
  - Research Site, Mykolaiv
  - Research Site, Odesa
  - Research Site, Poltava
  - Research Site, Uzhhorod
  - Research Site, Vinnytsia
  - Research Site, Zaporizhzhia
  - Research Site, Zhytomyr
- United Kingdom (20):
  - Research Site, Airdrie
  - Research Site, Bournemouth
  - Research Site, Cardiff
  - Research Site, Chelmsford
  - Research Site, Chorley
  - Research Site, East Kilbride
  - Research Site, Edgbaston
  - Research Site, Edinburgh
  - Research Site, Exeter
  - Research Site, Glasgow
  - Research Site, Hexham
  - Research Site, Leicester
  - Research Site, Liverpool
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Reading
  - Research Site, Romford
  - Research Site, Stevenage
  - Research Site, Swansea
  - Research Site, Torquay

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Nissen SE, Lincoff AM, Wolski K, Ballantyne CM, Kastelein JJP, Ridker PM, Ray KK, McGuire DK, Mozaffarian D, Koenig W, Davidson MH, Garcia M, Katona BG, Himmelmann A, Loss LE, Poole M, Menon V, Nicholls SJ. Association Between Achieved omega-3 Fatty Acid Levels and Major Adverse Cardiovascular Outcomes in Patients With High Cardiovascular Risk: A Secondary Analysis of the STRENGTH Trial. JAMA Cardiol. 2021 Aug 1;6(8):910-917. doi: 10.1001/jamacardio.2021.1157. PMID 33993205
- [Derived] Nicholls SJ, Lincoff AM, Garcia M, Bash D, Ballantyne CM, Barter PJ, Davidson MH, Kastelein JJP, Koenig W, McGuire DK, Mozaffarian D, Ridker PM, Ray KK, Katona BG, Himmelmann A, Loss LE, Rensfeldt M, Lundstrom T, Agrawal R, Menon V, Wolski K, Nissen SE. Effect of High-Dose Omega-3 Fatty Acids vs Corn Oil on Major Adverse Cardiovascular Events in Patients at High Cardiovascular Risk: The STRENGTH Randomized Clinical Trial. JAMA. 2020 Dec 8;324(22):2268-2280. doi: 10.1001/jama.2020.22258. PMID 33190147
- See also: redacted CSP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5881C00004&attachmentIdentifier=be55f883-e635-4760-b404-758aa7dd6106&fileName=redacted_CSP.pdf&versionIdentifier=
- See also: redacted SAP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5881C00004&attachmentIdentifier=5b7552b6-b71b-4a3b-8abf-513efc223986&fileName=redacted_SAP.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 686 study sites in 22 countries randomized subjects. The first patient was enrolled on 30 October 2014 and randomized on 11 November 2014. The last patient was randomized on 12 July 2017.
Groups:
- Epanova: Omega-3 carboxylic acid 4 x 1 gram capsule
- Placebo: Corn oil 4 x 1 gram capsule
Period: Overall Study
Arm/Group | Epanova | Placebo
Started | 6539 | 6539
Completed | 80 | 92
Not Completed | 6459 | 6447
Not completed — Death | 363 | 330
Not completed — Lost to Follow-up | 3 | 2
Not completed — Protocol Violation | 0 | 1
Not completed — Study terminated by sponsor | 5854 | 5901
Not completed — Withdrawal by Subject | 111 | 78
Not completed — Other reasons | 128 | 135

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Epanova | Placebo | Total
Number analyzed (Participants) | 6539 | 6539 | 13078
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.5 (8.98) | 62.5 (8.98) | 62.5 (8.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2289 | 2279 | 4568
  Male | 4250 | 4260 | 8510
Race/Ethnicity, Customized [Number; unit: Participants]
  WHITE | 5341 | 5382 | 10723
  BLACK OR AFRICAN AMERICAN | 180 | 166 | 346
  ASIAN | 698 | 657 | 1355
  NATIVE HAWAIIAN OR OTHER PACIFIC ISLANDER | 10 | 11 | 21
  AMERICAN INDIAN OR ALASKA NATIVE | 114 | 112 | 226
  OTHER | 159 | 154 | 313
  MULTIPLE | 33 | 47 | 80
  UNKNOWN | 4 | 10 | 14
  NOT REPORTED | 0 | 0 | 0
Region of Enrollment [Number; unit: Participants]
  Australia | 58 | 54 | 112
  Belgium | 53 | 51 | 104
  Canada | 187 | 177 | 364
  China | 357 | 356 | 713
  Czech Republic | 120 | 108 | 228
  Denmark | 48 | 73 | 121
  Estonia | 57 | 53 | 110
  Hungary | 561 | 562 | 1123
  Italy | 33 | 34 | 67
  Japan | 166 | 139 | 305
  Korea, Republic Of | 68 | 65 | 133
  Lithuania | 170 | 193 | 363
  Mexico | 152 | 155 | 307
  Netherlands | 206 | 215 | 421
  New Zealand | 74 | 77 | 151
  Poland | 501 | 492 | 993
  Russia | 307 | 326 | 633
  South Africa | 471 | 490 | 961
  Taiwan, Province Of China | 28 | 31 | 59
  Ukraine | 1009 | 955 | 1964
  United Kingdom | 377 | 382 | 759
  USA | 1536 | 1551 | 3087

OUTCOME MEASURES:

1. Primary Outcome: The Composite of Major Adverse Cardiovascular Events (MACE)
Description: MACE components include: cardiovascular (CV) death, nonfatal myocardial infarction (MI), nonfatal stroke, emergent/elective coronary revascularization, or hospitalization for unstable angina. Participants with no observed events are censored at the earliest of withdrawal of consent date and last study contact (defined as the latest of the dates of assessments contributing to an opportunity to assess as to whether the participant has had every component of the endpoint being analyzed).
Time Frame: From the date of randomization and up to completion of the end-of-treatment visit (Month 60) or at study closure
Population: Full Analysis Set
Measure: Number; unit: Number of Participants
Arm/Group | Epanova | Placebo
Number analyzed (Participants) | 6539 | 6539
Number of Participants | 785 | 795
Statistical Analysis 1: Comparison: Epanova vs Placebo; Test type: Superiority; p = 0.837, Regression, Cox — The hypothesis is tested at the 5% level. A hierarchical test sequence is used to address the issue of multiple testing; Hazard Ratio (HR) = 0.99, 95% CI 2-sided [0.90 to 1.09]

2. Secondary Outcome: The Composite of MACE in the Subgroup of Participants With Established CV Disease(CVD) at Baseline
Description: as for outcome 1
Time Frame: From the date of randomization and up to completion of the end-of-treatment visit (Month 60) or at study closure
Population: Full Analysis Set
Measure: Number; unit: Number of Participants
Arm/Group | Epanova | Placebo
Number analyzed (Participants) | 6539 | 6539
Number of Participants
  Overall number of participants | 785 | 795
  Number of participants with established cardiovascular disease (CVD) at baseline: number analyzed (Participants) | 3638 | 3678
  Number of participants with established cardiovascular disease (CVD) at baseline | 569 | 610
Statistical Analysis 1: Comparison: Epanova vs Placebo; Test type: Superiority; p = 0.269, Regression, Cox — The hypothesis is tested at the 5% level. A hierarchical test sequence is used to address the issue of multiple testing; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.84 to 1.05]

3. Secondary Outcome: The Composite of CV Events
Description: CV events include: cardiovascular (CV) death, non-fatal myocardial infarction (MI) and non-fatal stroke. Participants with no observed events are censored at the earliest of withdrawal of consent date and last study contact (defined as the latest of the dates of assessments contributing to an opportunity to assess as to whether the participant has had every component of the endpoint being analyzed).
Time Frame: From the date of randomization and up to completion of the end-of-treatment visit (Month 60) or at study closure
Population: Full Analysis Set
Measure: Number; unit: Number of Participants
Arm/Group | Epanova | Placebo
Number analyzed (Participants) | 6539 | 6539
Number of Participants | 541 | 517
Statistical Analysis 1: Comparison: Epanova vs Placebo; Test type: Superiority; p = 0.402, Regression, Cox — The hypothesis is tested at the 5% level. A hierarchical test sequence is used to address the issue of multiple testing; Hazard Ratio (HR) = 1.05, 95% CI 2-sided [0.93 to 1.19]

4. Secondary Outcome: The Composite of CV Events in the Subgroup of Participants With Established CV Disease (CVD) at Baseline
Description: as for outcome 3
Time Frame: From the date of randomization and up to completion of the end-of-treatment visit (Month 60) or at study closure
Population: Full Analysis Set
Measure: Number; unit: Number of Participants
Arm/Group | Epanova | Placebo
Number analyzed (Participants) | 6539 | 6539
Number of Participants
  Overall number of participants | 541 | 517
  Number of participants with established CVD at baseline: number analyzed (Participants) | 3638 | 3678
  Number of participants with established CVD at baseline | 383 | 385
Statistical Analysis 1: Comparison: Epanova vs Placebo; Test type: Superiority; p = 0.940, Regression, Cox — The hypothesis is tested at the 5% level. A hierarchical test sequence is used to address the issue of multiple testing; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.87 to 1.16]

5. Secondary Outcome: The Composite of Coronary Events
Description: Coronary events include: cardiac death (including death due to acute myocardial infarction, sudden cardiac death and death due to cardiovascular procedures), non-fatal myocardial infarction (MI), emergent/elective coronary revascularization and hospitalization for unstable angina. Participants with no observed events are censored at the earliest of withdrawal of consent date and last study contact (defined as the latest of the dates of assessments contributing to an opportunity to assess as to whether the participant has had every component of the endpoint being analyzed).
Time Frame: From the date of randomization and up to completion of the end-of-treatment visit (Month 60) or at study closure
Population: Full Analysis Set
Measure: Number; unit: Number of Participants
Arm/Group | Epanova | Placebo
Number analyzed (Participants) | 6539 | 6539
Number of Participants | 556 | 616
Statistical Analysis 1: Comparison: Epanova vs Placebo; Test type: Superiority; p = 0.092, Regression, Cox — The hypothesis is tested at the 5% level. A hierarchical test sequence is used to address the issue of multiple testing; Hazard Ratio (HR) = 0.91, 95% CI 2-sided [0.81 to 1.02]

6. Secondary Outcome: The Composite of Coronary Events in the Subgroup of Participants With Established CVD at Baseline
Description: Coronary events include: cardiac death (including death due to acute myocardial infarction, sudden cardiac death and death due to cardiovascular procedures), non-fatal myocardial infarction (MI), emergent/elective coronary revascularization and hospitalization for unstable angina. Participants with no observed events are censored at the earliest of withdrawal of consent date and last study contact (defined as the latest of the dates of assessments contributing to an opportunity to assess as to whether the participant has had every component of the endpoint being analyzed) in the subgroup of participants with established CVD at baseline
Time Frame: From the date of randomization and up to completion of the end-of-treatment visit (Month 60) or at study closure
Population: Full Analysis Set
Measure: Number; unit: Number of Participants
Arm/Group | Epanova | Placebo
Number analyzed (Participants) | 6539 | 6539
Number of Participants
  Overall number of participants | 556 | 616
  Number of participants with established CVD at baseline: number analyzed (Participants) | 3638 | 3678
  Number of participants with established CVD at baseline | 417 | 493
Statistical Analysis 1: Comparison: Epanova vs Placebo; Test type: Superiority; p = 0.016, Regression, Cox — The hypothesis is tested at the 5% level. A hierarchical test sequence is used to address the issue of multiple testing; Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.75 to 0.97]

7. Secondary Outcome: CV Death
Description: Participants with no observed events are censored at the latest of the date of last study contact (defined as the latest of the dates of assessments contributing to an opportunity to assess as to whether the participant has had every component of the endpoint being analyzed), last date known to be alive, and date of non-cardiovascular death.
Time Frame: From the date of randomization and up to completion of the end-of-treatment visit (Month 60) or at study closure
Measure: Number; unit: Number of Participants
Arm/Group | Epanova | Placebo
Number analyzed (Participants) | 6539 | 6539
Number of Participants | 228 | 211
Statistical Analysis 1: Comparison: Epanova vs Placebo; Test type: Superiority; p = 0.372, Regression, Cox — The hypothesis is tested at the 5% level. A hierarchical test sequence is used to address the issue of multiple testing; Hazard Ratio (HR) = 1.09, 95% CI 2-sided [0.90 to 1.31]

8. Secondary Outcome: CV Death in the Subgroup of Participants With Established CVD at Baseline
Description: Participants with no observed events are censored at the latest of the date of last study contact (defined as the latest of the dates of assessments contributing to an opportunity to assess as to whether the participant has had every component of the endpoint being analyzed), last date known to be alive, and date of non-cardiovascular death in the subgroup of participants with established CVD at baseline
Time Frame: From the date of randomization and up to completion of the end-of-treatment visit (Month 60) or at study closure
Population: Full Analysis Set
Measure: Number; unit: Number of Participants
Arm/Group | Epanova | Placebo
Number analyzed (Participants) | 6539 | 6539
Number of Participants
  Overall number of participants | 228 | 211
  Number of participants with established CVD at baseline: number analyzed (Participants) | 3638 | 3678
  Number of participants with established CVD at baseline | 152 | 138
Statistical Analysis 1: Comparison: Epanova vs Placebo; Test type: Superiority; p = 0.336, Regression, Cox — The hypothesis is tested at the 5% level. A hierarchical test sequence is used to address the issue of multiple testing; Hazard Ratio (HR) = 1.12, 95% CI 2-sided [0.89 to 1.41]

9. Secondary Outcome: All-cause Death
Description: Participants with no observed events are censored at the latest of the date of last study contact (defined as the latest of the dates of assessments contributing to an opportunity to assess as to whether the participant has had every component of the endpoint being analyzed) and last date known to be alive.
Time Frame: From the date of randomization and up to completion of the end-of-treatment visit (Month 60) or at study closure
Population: Full Analysis Set
Measure: Number; unit: Number of Participants
Arm/Group | Epanova | Placebo
Number analyzed (Participants) | 6539 | 6539
Number of Participants | 373 | 333
Statistical Analysis 1: Comparison: Epanova vs Placebo; Test type: Superiority; p = 0.112, Regression, Cox — The hypothesis is tested at the 5% level. A hierarchical test sequence is used to address the issue of multiple testing; Hazard Ratio (HR) = 1.13, 95% CI 2-sided [0.97 to 1.31]

10. Secondary Outcome: All-cause Death in the Subgroup of Participants With Established CVD at Baseline
Description: Participants with no observed events are censored at the latest of the date of last study contact (defined as the latest of the dates of assessments contributing to an opportunity to assess as to whether the participant has had every component of the endpoint being analyzed) and last date known to be alive in the subgroup of participants with established CVD at baseline
Time Frame: From the date of randomization and up to completion of the end-of-treatment visit (Month 60) or at study closure
Population: Full Analysis Set
Measure: Number; unit: Number of Participants
Arm/Group | Epanova | Placebo
Number analyzed (Participants) | 6539 | 6539
Number of Participants
  Overall number of participants | 373 | 333
  Number of participants with established CVD at baselne: number analyzed (Participants) | 3638 | 3678
  Number of participants with established CVD at baselne | 234 | 202
Statistical Analysis 1: Comparison: Epanova vs Placebo; Test type: Superiority; p = 0.091, Regression, Cox — The hypothesis is tested at the 5% level. A hierarchical test sequence is used to address the issue of multiple testing; Hazard Ratio (HR) = 1.18, 95% CI 2-sided [0.97 to 1.42]

11. Other Pre Specified Outcome: Emergent/Elective Coronary Revascularization
Description: Participants with no observed events are censored at the earliest of withdrawal of consent date and last study contact (defined as the latest of the dates of assessments contributing to an opportunity to assess as to whether the participant has had every component of the endpoint being analyzed).
Time Frame: From the date of randomization and up to completion of the end-of-treatment visit (Month 60) or at study closure
Population: Full Analysis Set
Measure: Number; unit: Number of Participants
Arm/Group | Epanova | Placebo
Number analyzed (Participants) | 6539 | 6539
Number of Participants | 414 | 441
Statistical Analysis 1: Comparison: Epanova vs Placebo; Test type: Superiority; p = 0.408, Regression, Cox — This endpoint was not in the testing sequence and therefore not under type I error control; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.83 to 1.08]

12. Other Pre Specified Outcome: Hospitalization for Unstable Angina
Description: as for outcome 11
Time Frame: From the date of randomization and up to completion of the end-of-treatment visit (Month 60) or at study closure
Population: Full Analysis Set
Measure: Number; unit: Number of Participants
Arm/Group | Epanova | Placebo
Number analyzed (Participants) | 6539 | 6539
Number of Participants | 87 | 104
Statistical Analysis 1: Comparison: Epanova vs Placebo; Test type: Superiority; p = 0.233, Regression, Cox — This endpoint was not in the testing sequence and therefore not under type I error control; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.63 to 1.12]

13. Other Pre Specified Outcome: Non-fatal Myocardial Infarction
Description: as for outcome 11
Time Frame: From the date of randomization and up to completion of the end-of-treatment visit (Month 60) or at study closure
Population: Full Analysis Set
Measure: Number; unit: Number of Participants
Arm/Group | Epanova | Placebo
Number analyzed (Participants) | 6539 | 6539
Number of Participants | 218 | 226
Statistical Analysis 1: Comparison: Epanova vs Placebo; Test type: Superiority; p = 0.770, Regression, Cox — This endpoint was not in the testing sequence and therefore not under type I error control; Hazard Ratio (HR) = 0.97, 95% CI 2-sided [0.81 to 1.17]

14. Other Pre Specified Outcome: Non-fatal Stroke
Description: as for outcome 11
Time Frame: From the date of randomization and up to completion of the end-of-treatment visit (Month 60) or at study closure
Population: Full Analysis Set
Measure: Number; unit: Number of Participants
Arm/Group | Epanova | Placebo
Number analyzed (Participants) | 6539 | 6539
Number of Participants | 142 | 125
Statistical Analysis 1: Comparison: Epanova vs Placebo; Test type: Superiority; p = 0.278, Regression, Cox — This endpoint was not in the testing sequence and therefore not under type I error control; Hazard Ratio (HR) = 1.14, 95% CI 2-sided [0.90 to 1.45]

ADVERSE EVENTS:
Time Frame: Predefined non-SAEs were collected from date of first IP dose until final visit/up to Month 60; if study treatment was discontinued prematurely, non-SAEs were recorded for ≤ 30 days after last IP dose. For AEs that are considered serious, lead to discontinuation, or result in dose modification, overdose, new onset diabetes mellitus, TIA, PHL cases or bleeding- related events were captured from date of first IP dose until final visit/up to Month 60, whether or not the participant discontinued IP.
Arm/Group | Epanova | Placebo
All-Cause Mortality (participants affected / at risk) | 373/6539 | 333/6539
Serious Adverse Events (participants affected / at risk) | 2259/6532 | 2195/6535
Other Adverse Events (participants affected / at risk) | 1405/6532 | 826/6535
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Epanova (N=6532) | Placebo (N=6535)
Agranulocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 15 (17) | 19 (25)
Anaemia macrocytic (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Antiphospholipid syndrome (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Blood loss anaemia (Blood and lymphatic system disorders) | 9 (9) | 6 (6)
Coagulopathy (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 9 (10) | 6 (6)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Microcytic anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Nephrogenic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Normocytic anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Polycythaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Splenic infarction (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Splenic thrombosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Splenomegaly (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3) | 3 (6)
Acute coronary syndrome (Cardiac disorders) | 13 (13) | 8 (8)
Acute left ventricular failure (Cardiac disorders) | 16 (16) | 8 (9)
Acute myocardial infarction (Cardiac disorders) | 40 (53) | 45 (47)
Adams-stokes syndrome (Cardiac disorders) | 0 (0) | 2 (2)
Angina pectoris (Cardiac disorders) | 92 (110) | 102 (113)
Angina unstable (Cardiac disorders) | 112 (125) | 141 (162)
Anginal equivalent (Cardiac disorders) | 1 (1) | 0 (0)
Aortic valve disease (Cardiac disorders) | 0 (0) | 2 (3)
Aortic valve incompetence (Cardiac disorders) | 1 (1) | 2 (2)
Aortic valve stenosis (Cardiac disorders) | 6 (8) | 3 (3)
Arrhythmia (Cardiac disorders) | 12 (12) | 5 (5)
Arteriosclerosis coronary artery (Cardiac disorders) | 19 (23) | 15 (20)
Arteriospasm coronary (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 150 (188) | 89 (103)
Atrial flutter (Cardiac disorders) | 14 (20) | 17 (20)
Atrial tachycardia (Cardiac disorders) | 2 (3) | 3 (5)
Atrioventricular block (Cardiac disorders) | 2 (2) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 7 (7) | 7 (7)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular block second degree (Cardiac disorders) | 4 (4) | 4 (4)
Atrioventricular dissociation (Cardiac disorders) | 1 (1) | 0 (0)
Bradyarrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 8 (8) | 9 (10)
Cardiac aneurysm (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 19 (19) | 11 (11)
Cardiac asthma (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac discomfort (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac disorder (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac failure (Cardiac disorders) | 90 (117) | 92 (132)
Cardiac failure acute (Cardiac disorders) | 27 (35) | 21 (25)
Cardiac failure chronic (Cardiac disorders) | 18 (21) | 21 (26)
Cardiac failure congestive (Cardiac disorders) | 60 (83) | 59 (77)
Cardiac tamponade (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac ventricular thrombosis (Cardiac disorders) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardio-respiratory distress (Cardiac disorders) | 0 (0) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 6 (6) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 9 (9) | 2 (2)
Cardiopulmonary failure (Cardiac disorders) | 3 (3) | 5 (5)
Cardiovascular deconditioning (Cardiac disorders) | 1 (1) | 0 (0)
Cardiovascular disorder (Cardiac disorders) | 0 (0) | 1 (1)
Cardiovascular insufficiency (Cardiac disorders) | 0 (0) | 1 (1)
Congestive cardiomyopathy (Cardiac disorders) | 2 (2) | 2 (2)
Coronary artery disease (Cardiac disorders) | 82 (89) | 61 (72)
Coronary artery insufficiency (Cardiac disorders) | 1 (1) | 1 (1)
Coronary artery occlusion (Cardiac disorders) | 3 (3) | 7 (8)
Coronary artery stenosis (Cardiac disorders) | 3 (3) | 8 (8)
Coronary artery thrombosis (Cardiac disorders) | 0 (0) | 2 (2)
Diastolic dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Extrasystoles (Cardiac disorders) | 1 (1) | 1 (1)
Hypertensive heart disease (Cardiac disorders) | 1 (1) | 0 (0)
Intracardiac thrombus (Cardiac disorders) | 1 (1) | 0 (0)
Ischaemic cardiomyopathy (Cardiac disorders) | 4 (5) | 10 (11)
Left ventricular dysfunction (Cardiac disorders) | 3 (3) | 4 (4)
Left ventricular failure (Cardiac disorders) | 6 (6) | 7 (7)
Metabolic cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Mitral valve disease (Cardiac disorders) | 0 (0) | 1 (2)
Mitral valve incompetence (Cardiac disorders) | 2 (2) | 4 (4)
Myocardial fibrosis (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 39 (43) | 51 (51)
Myocardial ischaemia (Cardiac disorders) | 27 (28) | 16 (17)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0)
Nodal arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Nodal rhythm (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Paroxysmal atrioventricular block (Cardiac disorders) | 1 (1) | 1 (1)
Pericardial effusion (Cardiac disorders) | 2 (2) | 3 (3)
Pericarditis (Cardiac disorders) | 1 (1) | 5 (5)
Pleuropericarditis (Cardiac disorders) | 0 (0) | 1 (1)
Postinfarction angina (Cardiac disorders) | 1 (1) | 0 (0)
Pulmonary valve stenosis (Cardiac disorders) | 0 (0) | 1 (2)
Pulseless electrical activity (Cardiac disorders) | 0 (0) | 4 (5)
Right ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
Silent myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Sinoatrial block (Cardiac disorders) | 0 (0) | 1 (1)
Sinus arrest (Cardiac disorders) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 3 (3) | 0 (0)
Sinus node dysfunction (Cardiac disorders) | 6 (6) | 5 (5)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 2 (2)
Supraventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 6 (6) | 5 (5)
Tachyarrhythmia (Cardiac disorders) | 0 (0) | 2 (2)
Tachycardia (Cardiac disorders) | 0 (0) | 3 (3)
Ventricular arrhythmia (Cardiac disorders) | 1 (1) | 1 (1)
Ventricular dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 5 (5) | 5 (5)
Ventricular fibrillation (Cardiac disorders) | 7 (8) | 8 (8)
Ventricular tachycardia (Cardiac disorders) | 13 (14) | 14 (16)
Arteriovenous malformation (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Atrial septal defect (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Cerebrovascular arteriovenous malformation (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Familial mediterranean fever (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Gastrointestinal arteriovenous malformation (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Hypertrophic cardiomyopathy (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Phimosis (Congenital, familial and genetic disorders) | 4 (4) | 1 (1)
Porokeratosis (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Pyloric stenosis (Congenital, familial and genetic disorders) | 1 (2) | 0 (0)
Deafness (Ear and labyrinth disorders) | 0 (0) | 2 (2)
Deafness neurosensory (Ear and labyrinth disorders) | 0 (0) | 2 (3)
Deafness unilateral (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Otolithiasis (Ear and labyrinth disorders) | 0 (0) | 2 (2)
Sudden hearing loss (Ear and labyrinth disorders) | 0 (0) | 1 (2)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 1 (2)
Vertigo (Ear and labyrinth disorders) | 12 (13) | 11 (11)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 2 (2)
Vestibular disorder (Ear and labyrinth disorders) | 1 (1) | 2 (2)
Acromegaly (Endocrine disorders) | 0 (0) | 1 (1)
Adrenal mass (Endocrine disorders) | 1 (1) | 1 (1)
Goitre (Endocrine disorders) | 4 (4) | 8 (8)
Hyperparathyroidism primary (Endocrine disorders) | 1 (1) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 2 (2) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 2 (2)
Parathyroid disorder (Endocrine disorders) | 0 (0) | 1 (1)
Thyroid mass (Endocrine disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 29 (35) | 20 (24)
Conjunctival erosion (Eye disorders) | 1 (1) | 0 (0)
Conjunctivochalasis (Eye disorders) | 1 (1) | 0 (0)
Corneal erosion (Eye disorders) | 1 (1) | 0 (0)
Dacryostenosis acquired (Eye disorders) | 1 (1) | 0 (0)
Diabetic retinopathy (Eye disorders) | 1 (1) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 1 (1)
Exophthalmos (Eye disorders) | 0 (0) | 1 (1)
Eyelid ptosis (Eye disorders) | 0 (0) | 2 (2)
Glaucoma (Eye disorders) | 4 (5) | 1 (1)
Iridocyclitis (Eye disorders) | 1 (1) | 0 (0)
Macular hole (Eye disorders) | 2 (2) | 0 (0)
Maculopathy (Eye disorders) | 1 (1) | 0 (0)
Open angle glaucoma (Eye disorders) | 2 (2) | 0 (0)
Optic ischaemic neuropathy (Eye disorders) | 1 (1) | 0 (0)
Retinal artery embolism (Eye disorders) | 2 (2) | 0 (0)
Retinal artery occlusion (Eye disorders) | 2 (2) | 1 (1)
Retinal detachment (Eye disorders) | 1 (1) | 2 (2)
Retinal haemorrhage (Eye disorders) | 1 (1) | 1 (1)
Retinal tear (Eye disorders) | 2 (2) | 0 (0)
Retinal vein occlusion (Eye disorders) | 1 (1) | 0 (0)
Retinopathy (Eye disorders) | 0 (0) | 1 (1)
Rhegmatogenous retinal detachment (Eye disorders) | 0 (0) | 1 (3)
Tractional retinal detachment (Eye disorders) | 0 (0) | 1 (2)
Vitreous detachment (Eye disorders) | 1 (1) | 0 (0)
Vitreous disorder (Eye disorders) | 1 (1) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 2 (2) | 1 (1)
Abdominal adhesions (Gastrointestinal disorders) | 1 (1) | 2 (2)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 5 (5) | 5 (5)
Abdominal hernia obstructive (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal incarcerated hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 8 (9) | 9 (11)
Abdominal pain lower (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 3 (3)
Abdominal wall haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Alcoholic pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anal fistula (Gastrointestinal disorders) | 2 (2) | 0 (0)
Anal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anogenital dysplasia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Barrett's oesophagus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chronic gastritis (Gastrointestinal disorders) | 3 (3) | 7 (8)
Coeliac artery stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 7 (7) | 7 (8)
Colitis ischaemic (Gastrointestinal disorders) | 3 (3) | 2 (2)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1) | 3 (4)
Colonic fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 6 (7) | 5 (5)
Crohn's disease (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dental cyst (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diabetic gastroparesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diabetic gastropathy (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diaphragmatic hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 21 (21) | 10 (11)
Dieulafoy's vascular malformation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diverticular perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diverticulum (Gastrointestinal disorders) | 3 (3) | 4 (4)
Diverticulum intestinal (Gastrointestinal disorders) | 3 (3) | 0 (0)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 (1) | 3 (3)
Duodenal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal polyp (Gastrointestinal disorders) | 1 (1) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 5 (5) | 3 (3)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 4 (4) | 3 (3)
Duodenal ulcer perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Duodenogastric reflux (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysbiosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 1 (1)
Enteritis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Enterovesical fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Erosive duodenitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Faecaloma (Gastrointestinal disorders) | 0 (0) | 2 (2)
Functional gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric polyps (Gastrointestinal disorders) | 3 (3) | 2 (2)
Gastric ulcer (Gastrointestinal disorders) | 5 (5) | 1 (1)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 4 (4) | 1 (1)
Gastric ulcer perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 9 (9) | 8 (8)
Gastritis erosive (Gastrointestinal disorders) | 6 (6) | 3 (3)
Gastritis haemorrhagic (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastroduodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastrointestinal erosion (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 24 (31) | 10 (11)
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrointestinal polyp haemorrhage (Gastrointestinal disorders) | 1 (1) | 2 (2)
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal vascular malformation haemorrhagic (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 7 (7) | 7 (7)
Gingival bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 2 (2) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 4 (4) | 1 (1)
Haemorrhagic erosive gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 2 (2) | 6 (7)
Haemorrhoids (Gastrointestinal disorders) | 5 (5) | 5 (5)
Haemorrhoids thrombosed (Gastrointestinal disorders) | 0 (0) | 3 (4)
Hiatus hernia (Gastrointestinal disorders) | 4 (4) | 1 (1)
Ileus (Gastrointestinal disorders) | 3 (3) | 1 (1)
Ileus paralytic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Incarcerated inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 18 (19) | 11 (12)
Intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Intestinal mass (Gastrointestinal disorders) | 1 (1) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 7 (7) | 4 (4)
Intestinal perforation (Gastrointestinal disorders) | 2 (3) | 0 (0)
Intestinal polyp (Gastrointestinal disorders) | 1 (1) | 3 (3)
Intestinal pseudo-obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 2 (2)
Large intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1)
Large intestinal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 14 (15) | 13 (19)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 2 (2)
Mechanical ileus (Gastrointestinal disorders) | 0 (0) | 2 (2)
Melaena (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mesenteric artery stenosis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Mesenteric haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mesenteric vascular insufficiency (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (4) | 3 (3)
Noninfective sialoadenitis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Obstructive pancreatitis (Gastrointestinal disorders) | 3 (3) | 0 (0)
Oedematous pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal achalasia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal spasm (Gastrointestinal disorders) | 1 (1) | 2 (2)
Oesophageal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 2 (2) | 1 (1)
Pancreatic disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 11 (11) | 10 (10)
Pancreatitis acute (Gastrointestinal disorders) | 12 (16) | 11 (11)
Pancreatitis chronic (Gastrointestinal disorders) | 0 (0) | 3 (3)
Peptic ulcer (Gastrointestinal disorders) | 0 (0) | 3 (3)
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pharyngo-oesophageal diverticulum (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pneumatosis intestinalis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 7 (8) | 5 (5)
Rectal polyp (Gastrointestinal disorders) | 0 (0) | 1 (2)
Rectal prolapse (Gastrointestinal disorders) | 1 (1) | 0 (0)
Reflux gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Retroperitoneal fibrosis (Gastrointestinal disorders) | 1 (3) | 0 (0)
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Retroperitoneal mass (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 5 (6) | 9 (12)
Thrombosis mesenteric vessel (Gastrointestinal disorders) | 1 (1) | 0 (0)
Tongue cyst (Gastrointestinal disorders) | 0 (0) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 5 (5) | 2 (2)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 12 (12) | 3 (3)
Volvulus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Volvulus of small bowel (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 8 (9) | 1 (1)
Adverse drug reaction (General disorders) | 1 (1) | 1 (1)
Adverse event (General disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 2 (2)
Cardiac death (General disorders) | 3 (3) | 3 (3)
Catheter site haemorrhage (General disorders) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 2 (2) | 4 (4)
Chest pain (General disorders) | 10 (10) | 23 (23)
Complication associated with device (General disorders) | 1 (1) | 1 (1)
Cyst (General disorders) | 0 (0) | 1 (1)
Death (General disorders) | 57 (57) | 38 (38)
Decreased activity (General disorders) | 0 (0) | 1 (1)
Device related thrombosis (General disorders) | 0 (0) | 1 (1)
Drowning (General disorders) | 0 (0) | 1 (1)
Drug intolerance (General disorders) | 1 (1) | 1 (1)
Exercise tolerance decreased (General disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 1 (1) | 1 (1)
General physical health deterioration (General disorders) | 2 (2) | 0 (0)
Generalised oedema (General disorders) | 0 (0) | 1 (1)
Hernia (General disorders) | 0 (0) | 1 (1)
Impaired healing (General disorders) | 0 (0) | 2 (2)
Implant site haematoma (General disorders) | 1 (1) | 0 (0)
Implant site inflammation (General disorders) | 1 (1) | 0 (0)
Inflammation (General disorders) | 1 (1) | 0 (0)
Injection site phlebitis (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 2 (2)
Medical device site haematoma (General disorders) | 0 (0) | 1 (1)
Mucosal inflammation (General disorders) | 1 (1) | 0 (0)
Multi-organ disorder (General disorders) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 5 (5) | 2 (2)
No adverse event (General disorders) | 1 (1) | 0 (0)
Nodule (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 51 (69) | 51 (53)
Oedema peripheral (General disorders) | 0 (0) | 3 (4)
Organ failure (General disorders) | 1 (1) | 0 (0)
Pelvic mass (General disorders) | 0 (0) | 1 (1)
Perforation (General disorders) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 2 (2) | 3 (3)
Pyrexia (General disorders) | 3 (3) | 4 (4)
Retention cyst (General disorders) | 1 (1) | 0 (0)
Stent-graft endoleak (General disorders) | 1 (1) | 1 (1)
Sudden cardiac death (General disorders) | 5 (5) | 4 (4)
Sudden death (General disorders) | 4 (4) | 3 (3)
Surgical failure (General disorders) | 1 (1) | 1 (1)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 1 (1)
Ulcer haemorrhage (General disorders) | 1 (1) | 0 (0)
Unevaluable event (General disorders) | 1 (1) | 0 (0)
Vascular stent occlusion (General disorders) | 1 (1) | 0 (0)
Vascular stent stenosis (General disorders) | 3 (3) | 2 (2)
Vascular stent thrombosis (General disorders) | 1 (1) | 5 (5)
Bile duct stenosis (Hepatobiliary disorders) | 1 (2) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 4 (6) | 3 (3)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Biliary tract disorder (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 6 (6) | 5 (5)
Cholangitis acute (Hepatobiliary disorders) | 2 (2) | 2 (2)
Cholecystitis (Hepatobiliary disorders) | 13 (13) | 17 (18)
Cholecystitis acute (Hepatobiliary disorders) | 20 (20) | 12 (13)
Cholecystitis chronic (Hepatobiliary disorders) | 4 (4) | 4 (5)
Cholelithiasis (Hepatobiliary disorders) | 27 (28) | 15 (16)
Chronic hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 3 (3) | 2 (2)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 2 (2)
Hepatic steatosis (Hepatobiliary disorders) | 1 (1) | 2 (2)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Ischaemic hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Jaundice (Hepatobiliary disorders) | 0 (0) | 1 (1)
Jaundice cholestatic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Liver disorder (Hepatobiliary disorders) | 0 (0) | 1 (1)
Non-alcoholic steatohepatitis (Hepatobiliary disorders) | 2 (2) | 1 (1)
Nonalcoholic fatty liver disease (Hepatobiliary disorders) | 2 (2) | 1 (1)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Post cholecystectomy syndrome (Hepatobiliary disorders) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 3 (3)
Anaphylactic shock (Immune system disorders) | 1 (1) | 1 (1)
Contrast media allergy (Immune system disorders) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 2 (2) | 1 (1)
Heart transplant rejection (Immune system disorders) | 0 (0) | 1 (2)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Kidney transplant rejection (Immune system disorders) | 1 (1) | 0 (0)
Sarcoidosis (Immune system disorders) | 0 (0) | 1 (1)
Abdominal abscess (Infections and infestations) | 2 (2) | 1 (1)
Abdominal wall abscess (Infections and infestations) | 2 (2) | 2 (3)
Abdominal wall infection (Infections and infestations) | 0 (0) | 1 (1)
Abscess (Infections and infestations) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 4 (4) | 6 (6)
Acarodermatitis (Infections and infestations) | 0 (0) | 1 (1)
Acquired immunodeficiency syndrome (Infections and infestations) | 0 (0) | 1 (1)
Acute hepatitis b (Infections and infestations) | 1 (1) | 0 (0)
Acute sinusitis (Infections and infestations) | 1 (1) | 3 (4)
Adenovirus infection (Infections and infestations) | 1 (1) | 1 (1)
Anal abscess (Infections and infestations) | 1 (1) | 3 (3)
Appendicitis (Infections and infestations) | 9 (9) | 14 (14)
Appendicitis perforated (Infections and infestations) | 5 (5) | 1 (1)
Arthritis bacterial (Infections and infestations) | 0 (0) | 4 (4)
Arthritis infective (Infections and infestations) | 2 (2) | 1 (1)
Atypical pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Bacteraemia (Infections and infestations) | 4 (4) | 4 (4)
Bacterial colitis (Infections and infestations) | 0 (0) | 1 (1)
Bacterial infection (Infections and infestations) | 1 (1) | 0 (0)
Bacterial prostatitis (Infections and infestations) | 0 (0) | 1 (1)
Beta haemolytic streptococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Biliary sepsis (Infections and infestations) | 1 (1) | 2 (2)
Borrelia infection (Infections and infestations) | 0 (0) | 1 (1)
Breast abscess (Infections and infestations) | 2 (2) | 1 (1)
Bronchitis (Infections and infestations) | 10 (11) | 23 (23)
Bronchitis viral (Infections and infestations) | 1 (1) | 3 (3)
Bursitis infective (Infections and infestations) | 0 (0) | 1 (1)
Campylobacter colitis (Infections and infestations) | 1 (1) | 1 (1)
Campylobacter gastroenteritis (Infections and infestations) | 2 (2) | 0 (0)
Candida pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Carbuncle (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 39 (46) | 46 (52)
Cellulitis of male external genital organ (Infections and infestations) | 2 (2) | 0 (0)
Cellulitis staphylococcal (Infections and infestations) | 1 (1) | 1 (1)
Chest wall abscess (Infections and infestations) | 1 (1) | 1 (1)
Cholangitis infective (Infections and infestations) | 1 (1) | 0 (0)
Cholecystitis infective (Infections and infestations) | 1 (1) | 3 (4)
Chronic sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 2 (2) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 4 (5) | 1 (1)
Dermatitis infected (Infections and infestations) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 2 (4) | 2 (2)
Diabetic foot infection (Infections and infestations) | 1 (1) | 3 (4)
Diabetic gangrene (Infections and infestations) | 1 (1) | 0 (0)
Diarrhoea infectious (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 13 (16) | 9 (12)
Diverticulitis intestinal haemorrhagic (Infections and infestations) | 1 (1) | 0 (0)
Dysentery (Infections and infestations) | 1 (1) | 0 (0)
Emphysematous pyelonephritis (Infections and infestations) | 1 (1) | 1 (1)
Empyema (Infections and infestations) | 0 (0) | 1 (1)
Endocarditis (Infections and infestations) | 1 (1) | 2 (2)
Endocarditis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Enterococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Epidemic pleurodynia (Infections and infestations) | 1 (1) | 0 (0)
Epididymitis (Infections and infestations) | 1 (2) | 0 (0)
Erysipelas (Infections and infestations) | 6 (10) | 6 (7)
Escherichia bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Escherichia infection (Infections and infestations) | 0 (0) | 1 (1)
Escherichia pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Escherichia sepsis (Infections and infestations) | 2 (2) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 2 (2)
External ear cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Extradural abscess (Infections and infestations) | 1 (1) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 1 (1)
Fournier's gangrene (Infections and infestations) | 1 (1) | 0 (0)
Fungal infection (Infections and infestations) | 1 (1) | 0 (0)
Gallbladder abscess (Infections and infestations) | 1 (1) | 0 (0)
Gallbladder empyema (Infections and infestations) | 1 (1) | 0 (0)
Gangrene (Infections and infestations) | 7 (7) | 9 (11)
Gastroenteritis (Infections and infestations) | 15 (16) | 20 (20)
Gastroenteritis clostridial (Infections and infestations) | 1 (1) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 4 (5) | 4 (4)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 1 (1)
Gastrointestinal viral infection (Infections and infestations) | 1 (1) | 1 (1)
Genitourinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Graft infection (Infections and infestations) | 1 (1) | 0 (0)
Groin abscess (Infections and infestations) | 3 (3) | 0 (0)
Hiv infection (Infections and infestations) | 1 (1) | 0 (0)
Haematoma infection (Infections and infestations) | 1 (1) | 0 (0)
Helicobacter gastritis (Infections and infestations) | 1 (1) | 0 (0)
Hepatic cyst infection (Infections and infestations) | 0 (0) | 1 (1)
Hepatitis c (Infections and infestations) | 0 (0) | 3 (3)
Herpes zoster (Infections and infestations) | 4 (4) | 4 (4)
Implant site infection (Infections and infestations) | 0 (0) | 2 (2)
Incision site cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Infected cyst (Infections and infestations) | 1 (1) | 0 (0)
Infected dermal cyst (Infections and infestations) | 1 (1) | 0 (0)
Infected skin ulcer (Infections and infestations) | 1 (1) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Infectious pleural effusion (Infections and infestations) | 1 (1) | 0 (0)
Infective aneurysm (Infections and infestations) | 0 (0) | 1 (1)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 2 (2) | 3 (3)
Infective tenosynovitis (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 12 (13) | 15 (15)
Intervertebral discitis (Infections and infestations) | 1 (1) | 0 (0)
Intestinal gangrene (Infections and infestations) | 0 (0) | 1 (1)
Kidney infection (Infections and infestations) | 0 (0) | 1 (1)
Klebsiella infection (Infections and infestations) | 0 (0) | 1 (1)
Large intestine infection (Infections and infestations) | 0 (0) | 1 (1)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1)
Liver abscess (Infections and infestations) | 3 (6) | 2 (2)
Localised infection (Infections and infestations) | 1 (1) | 5 (9)
Lower respiratory tract infection (Infections and infestations) | 8 (8) | 12 (13)
Lower respiratory tract infection bacterial (Infections and infestations) | 1 (1) | 0 (0)
Lyme disease (Infections and infestations) | 2 (2) | 0 (0)
Lymphangitis (Infections and infestations) | 0 (0) | 1 (1)
Mastitis (Infections and infestations) | 0 (0) | 1 (1)
Mediastinitis (Infections and infestations) | 2 (2) | 0 (0)
Medical device site abscess (Infections and infestations) | 0 (0) | 1 (1)
Medical device site infection (Infections and infestations) | 1 (1) | 1 (1)
Medical device site joint infection (Infections and infestations) | 1 (1) | 0 (0)
Meningitis (Infections and infestations) | 0 (0) | 1 (1)
Meningitis bacterial (Infections and infestations) | 0 (0) | 2 (3)
Meningoencephalitis herpetic (Infections and infestations) | 1 (1) | 0 (0)
Moraxella infection (Infections and infestations) | 0 (0) | 1 (1)
Mycetoma mycotic (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Necrotising fasciitis (Infections and infestations) | 2 (2) | 0 (0)
Oesophageal candidiasis (Infections and infestations) | 2 (2) | 1 (1)
Orchitis (Infections and infestations) | 1 (1) | 1 (1)
Osteomyelitis (Infections and infestations) | 9 (11) | 12 (16)
Osteomyelitis acute (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis chronic (Infections and infestations) | 0 (0) | 1 (1)
Otitis externa (Infections and infestations) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 1 (1) | 1 (1)
Otitis media acute (Infections and infestations) | 2 (2) | 0 (0)
Otitis media bacterial (Infections and infestations) | 0 (0) | 1 (1)
Otitis media chronic (Infections and infestations) | 0 (0) | 1 (1)
Parainfluenzae virus infection (Infections and infestations) | 0 (0) | 1 (1)
Parotitis (Infections and infestations) | 0 (0) | 2 (2)
Pelvic infection (Infections and infestations) | 0 (0) | 1 (1)
Perineal abscess (Infections and infestations) | 0 (0) | 1 (1)
Periodontitis (Infections and infestations) | 0 (0) | 1 (1)
Perirectal abscess (Infections and infestations) | 2 (2) | 0 (0)
Peritonitis (Infections and infestations) | 1 (1) | 3 (3)
Peritonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Pilonidal cyst (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 113 (130) | 126 (135)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 2 (2)
Pneumonia haemophilus (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia legionella (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia pseudomonal (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia staphylococcal (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia streptococcal (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia viral (Infections and infestations) | 2 (2) | 0 (0)
Post procedural cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Post procedural sepsis (Infections and infestations) | 4 (4) | 1 (1)
Postoperative abscess (Infections and infestations) | 2 (2) | 0 (0)
Postoperative wound infection (Infections and infestations) | 8 (8) | 2 (2)
Pseudomonas infection (Infections and infestations) | 1 (1) | 0 (0)
Psoas abscess (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary nocardiosis (Infections and infestations) | 0 (0) | 1 (1)
Pulmonary sepsis (Infections and infestations) | 1 (1) | 1 (1)
Pyelonephritis (Infections and infestations) | 9 (9) | 12 (12)
Pyelonephritis acute (Infections and infestations) | 7 (9) | 3 (3)
Pyelonephritis chronic (Infections and infestations) | 5 (5) | 1 (1)
Rectal abscess (Infections and infestations) | 1 (1) | 0 (0)
Renal abscess (Infections and infestations) | 1 (1) | 0 (0)
Renal cyst infection (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1)
Rotavirus infection (Infections and infestations) | 0 (0) | 1 (1)
Salmonellosis (Infections and infestations) | 1 (1) | 0 (0)
Scrotal abscess (Infections and infestations) | 0 (0) | 2 (2)
Sepsis (Infections and infestations) | 49 (51) | 43 (47)
Septic necrosis (Infections and infestations) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 8 (8) | 7 (10)
Sinobronchitis (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 2 (2) | 2 (2)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal abscess (Infections and infestations) | 0 (0) | 2 (2)
Staphylococcal bacteraemia (Infections and infestations) | 2 (2) | 3 (3)
Staphylococcal infection (Infections and infestations) | 1 (1) | 3 (3)
Staphylococcal sepsis (Infections and infestations) | 1 (1) | 4 (4)
Streptococcal abscess (Infections and infestations) | 1 (1) | 0 (0)
Streptococcal sepsis (Infections and infestations) | 2 (2) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 2 (2)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 1 (1) | 1 (1)
Tracheitis (Infections and infestations) | 0 (0) | 1 (1)
Tracheobronchitis (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 3 (3)
Urinary tract infection (Infections and infestations) | 24 (26) | 36 (40)
Urosepsis (Infections and infestations) | 9 (9) | 9 (9)
Vestibular neuronitis (Infections and infestations) | 3 (4) | 2 (2)
Viral infection (Infections and infestations) | 1 (1) | 2 (2)
Wound infection (Infections and infestations) | 1 (1) | 7 (7)
Wound infection bacterial (Infections and infestations) | 1 (1) | 0 (0)
Wound sepsis (Infections and infestations) | 2 (2) | 1 (1)
Abdominal injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Acetabulum fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Airway complication of anaesthesia (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Animal bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 5 (5) | 9 (10)
Arterial bypass occlusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Arterial bypass stenosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Back injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Bone contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Brain contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Burns second degree (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Carotid artery restenosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Chest injury (Injury, poisoning and procedural complications) | 0 (0) | 5 (5)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 1 (3) | 0 (0)
Coronary artery restenosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Cystitis radiation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Epicondylitis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Eyelid injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 15 (19) | 10 (10)
Femoral neck fracture (Injury, poisoning and procedural complications) | 9 (9) | 7 (7)
Femur fracture (Injury, poisoning and procedural complications) | 8 (8) | 9 (9)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Foot fracture (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Forearm fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Foreign body aspiration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Foreign body in gastrointestinal tract (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Fracture displacement (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Frostbite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 5 (5) | 8 (8)
Hip fracture (Injury, poisoning and procedural complications) | 4 (4) | 11 (11)
Humerus fracture (Injury, poisoning and procedural complications) | 5 (5) | 6 (6)
Hyphaema (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Incisional hernia (Injury, poisoning and procedural complications) | 5 (5) | 4 (5)
Inflammation of wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Intentional overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 4 (4)
Joint injury (Injury, poisoning and procedural complications) | 1 (2) | 3 (3)
Ligament rupture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Limb injury (Injury, poisoning and procedural complications) | 2 (2) | 3 (4)
Limb traumatic amputation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 3 (4) | 3 (3)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Mallet finger (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 4 (4) | 3 (3)
Multiple fractures (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Multiple injuries (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Muscle injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Muscle rupture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Neck injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Patella fracture (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Pelvic organ injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Peripheral artery restenosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Peripheral nerve injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Periprosthetic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pharyngeal contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post concussion syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post laminectomy syndrome (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural complication (Injury, poisoning and procedural complications) | 2 (2) | 2 (3)
Post procedural fever (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 4 (4)
Post procedural haematuria (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 7 (8) | 7 (7)
Post procedural swelling (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative delirium (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative hypotension (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Postoperative ileus (Injury, poisoning and procedural complications) | 2 (2) | 2 (5)
Postoperative respiratory failure (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural hypotension (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural nausea (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 7 (7)
Pseudomeningocele (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pubis fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pulmonary contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radiation dysphagia (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radiation injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 6 (6)
Rib fracture (Injury, poisoning and procedural complications) | 7 (7) | 5 (5)
Road traffic accident (Injury, poisoning and procedural complications) | 6 (6) | 5 (5)
Scapula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Shunt thrombosis (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Skeletal injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Skin laceration (Injury, poisoning and procedural complications) | 2 (2) | 6 (6)
Skull fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skull fractured base (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Soft tissue injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Spinal compression fracture (Injury, poisoning and procedural complications) | 9 (10) | 5 (5)
Spinal cord injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Splenic injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Splenic rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Stress fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 11 (14) | 9 (10)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Suture related complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tendon injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 6 (6) | 5 (5)
Thermal burn (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Toxicity to various agents (Injury, poisoning and procedural complications) | 2 (2) | 5 (5)
Traumatic arthrosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic haemothorax (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic ulcer (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ulna fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Urethral injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular graft occlusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Vascular procedure complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Wound (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Anticoagulation drug level above therapeutic (Investigations) | 2 (2) | 0 (0)
Anticoagulation drug level increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Blood calcium decreased (Investigations) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Blood glucose abnormal (Investigations) | 3 (3) | 0 (0)
Blood glucose decreased (Investigations) | 1 (1) | 1 (1)
Blood glucose fluctuation (Investigations) | 0 (0) | 1 (2)
Blood glucose increased (Investigations) | 1 (1) | 2 (2)
Blood lactic acid increased (Investigations) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 0 (0) | 3 (3)
C-reactive protein increased (Investigations) | 1 (1) | 0 (0)
Ejection fraction decreased (Investigations) | 1 (1) | 0 (0)
Electrocardiogram change (Investigations) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1)
Glycosylated haemoglobin increased (Investigations) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0)
Heart rate irregular (Investigations) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0)
International normalised ratio increased (Investigations) | 1 (1) | 0 (0)
Intraocular pressure increased (Investigations) | 1 (1) | 0 (0)
Liver function test abnormal (Investigations) | 0 (0) | 1 (1)
Liver function test increased (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
Prostatic specific antigen increased (Investigations) | 1 (1) | 0 (0)
Sinus rhythm (Investigations) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 1 (1) | 1 (1)
Transplant evaluation (Investigations) | 0 (0) | 1 (1)
Trial of void (Investigations) | 0 (0) | 1 (1)
Troponin i increased (Investigations) | 0 (0) | 2 (2)
Troponin increased (Investigations) | 2 (2) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0)
Weight increased (Investigations) | 1 (1) | 0 (0)
Cardiometabolic syndrome (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Central obesity (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 8 (9) | 12 (13)
Diabetes mellitus (Metabolism and nutrition disorders) | 43 (47) | 49 (50)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 26 (29) | 24 (32)
Diabetic complication (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 6 (6) | 6 (6)
Diabetic ketosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 16 (16) | 13 (14)
Electrolyte imbalance (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 3 (3) | 3 (3)
Gout (Metabolism and nutrition disorders) | 6 (6) | 7 (9)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 13 (13) | 12 (14)
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperhomocysteinaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 5 (5) | 13 (13)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Hypervolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (3)
Hypoglycaemia (Metabolism and nutrition disorders) | 14 (15) | 16 (18)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 3 (4)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hyponatraemia (Metabolism and nutrition disorders) | 4 (4) | 1 (1)
Hypovolaemia (Metabolism and nutrition disorders) | 4 (4) | 1 (1)
Ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Lactic acidosis (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 6 (6) | 10 (10)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 28 (32) | 18 (19)
Vitamin b12 deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 (11) | 12 (14)
Arthritis (Musculoskeletal and connective tissue disorders) | 8 (8) | 6 (6)
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (10) | 11 (11)
Bone lesion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 6 (6) | 4 (4)
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Costochondritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Crystal arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Foot deformity (Musculoskeletal and connective tissue disorders) | 4 (5) | 0 (0)
Fracture nonunion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Inguinal mass (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Intervertebral disc displacement (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 13 (13) | 17 (17)
Joint ankylosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Limb deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Limb mass (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 18 (18) | 11 (11)
Mandibular mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Meniscal degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 7 (7) | 9 (9)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 6 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Myopathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Osteitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 66 (69) | 58 (67)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (6) | 4 (4)
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 (3) | 2 (2)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Rheumatic disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 6 (6) | 10 (10)
Spinal instability (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 17 (17) | 8 (8)
Spinal pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 4 (4) | 11 (11)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (3)
Spondylolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tendon disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Thoracic spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Acoustic neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Acute promyelocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (5) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (5) | 6 (6)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 0 (0)
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Angiomyolipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
B-cell prolymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
B-cell small lymphocytic lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 15 (15) | 17 (22)
Benign bone neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Benign neoplasm of adrenal gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign neoplasm of bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign neoplasm of eyelid (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Benign ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Benign pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 (9) | 9 (10)
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Bladder cancer stage i, with cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 6 (7)
Bladder squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 5 (5)
Bladder transitional cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Bone cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3)
Brain cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 (9) | 17 (17)
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 3 (3)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Breast cancer stage i (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer stage ii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (4)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Bronchioloalveolar carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Carcinoid tumour pulmonary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Cardiac neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Castleman's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (4) | 4 (4)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 (11) | 20 (21)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Colon cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon cancer stage iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 0 (0)
Colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Colorectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Craniopharyngioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Diffuse large b-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ear neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Essential thrombocythaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Female reproductive neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastric adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 4 (4)
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Haemangioma of bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Head and neck cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 5 (5)
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 3 (3)
Immune reconstitution inflammatory syndrome associated kaposi's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Intestinal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Intraductal papillary mucinous neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Intraductal papilloma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 5 (5)
Keratinising squamous cell carcinoma of nasopharynx (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Large intestine benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (4)
Laryngeal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Lentigo maligna (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (9) | 9 (11)
Lung adenocarcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (4) | 2 (2)
Lung carcinoma cell type unspecified stage ii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung carcinoma cell type unspecified stage iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 3 (3)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 (8) | 12 (12)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11 (12) | 7 (7)
Malignant melanoma stage iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant neoplasm of eye (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant neoplasm of renal pelvis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant neoplasm of spinal cord (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant polyp (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Mantle cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 2 (2)
Meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 0 (0)
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Metastases to pleura (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to rectum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to soft tissue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Metastatic uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Mucoepidermoid carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Myelofibrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 4 (4)
Neoplasm of appendix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neoplasm prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Neuroendocrine carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Neuroendocrine carcinoma of the skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Nodular melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Non-hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3)
Non-hodgkin's lymphoma stage i (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 4 (4)
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Non-small cell lung cancer stage iiia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Non-small cell lung cancer stage iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1)
Oesophageal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 2 (2)
Oesophageal papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Oesophageal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
Oral neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oropharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oropharyngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ovarian endometrioid carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ovarian granulosa cell tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Paget's disease of the vulva (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 12 (12) | 4 (6)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 2 (2)
Pancreatic carcinoma stage iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Papillary renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3)
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 4 (6)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 4 (5)
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 34 (34) | 33 (34)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (4)
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer stage iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Queyrat erythroplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 4 (4)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 4 (4)
Rectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Rectal cancer stage iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rectosigmoid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal cancer stage i (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (7) | 0 (0)
Renal cell carcinoma stage iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Retroperitoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Salivary gland adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Schwannoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Secretory adenoma of pituitary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Sinonasal papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Small intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Soft tissue neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Spindle cell sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (4) | 4 (5)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 5 (5)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 8 (10)
Squamous cell carcinoma of the oral cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3)
Superficial spreading melanoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3)
Thyroid cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tongue neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 4 (4)
Ureteric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Urinary tract neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 5 (5)
Vaginal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Altered state of consciousness (Nervous system disorders) | 2 (2) | 1 (1)
Amnesia (Nervous system disorders) | 1 (1) | 1 (1)
Amyotrophic lateral sclerosis (Nervous system disorders) | 1 (2) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 2 (2)
Autonomic nervous system imbalance (Nervous system disorders) | 1 (1) | 0 (0)
Balance disorder (Nervous system disorders) | 0 (0) | 1 (1)
Basal ganglia infarction (Nervous system disorders) | 1 (1) | 0 (0)
Basilar artery aneurysm (Nervous system disorders) | 1 (1) | 0 (0)
Basilar artery stenosis (Nervous system disorders) | 1 (1) | 0 (0)
Brain stem ischaemia (Nervous system disorders) | 1 (1) | 0 (0)
Brain stem stroke (Nervous system disorders) | 0 (0) | 1 (1)
Carotid arteriosclerosis (Nervous system disorders) | 1 (1) | 2 (2)
Carotid artery disease (Nervous system disorders) | 2 (2) | 0 (0)
Carotid artery occlusion (Nervous system disorders) | 1 (1) | 2 (2)
Carotid artery stenosis (Nervous system disorders) | 17 (18) | 14 (15)
Carpal tunnel syndrome (Nervous system disorders) | 3 (3) | 4 (4)
Cerebellar infarction (Nervous system disorders) | 0 (0) | 2 (2)
Cerebellar stroke (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral artery stenosis (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral haematoma (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 2 (2) | 2 (2)
Cerebral infarction (Nervous system disorders) | 12 (12) | 17 (18)
Cerebral ischaemia (Nervous system disorders) | 6 (6) | 12 (15)
Cerebral small vessel ischaemic disease (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral venous sinus thrombosis (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 45 (46) | 42 (43)
Cerebrovascular insufficiency (Nervous system disorders) | 4 (4) | 4 (4)
Cerebrovascular stenosis (Nervous system disorders) | 1 (1) | 0 (0)
Cervical radiculopathy (Nervous system disorders) | 1 (1) | 2 (2)
Cervicobrachial syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Cluster headache (Nervous system disorders) | 1 (1) | 0 (0)
Cognitive disorder (Nervous system disorders) | 0 (0) | 1 (1)
Dementia (Nervous system disorders) | 4 (4) | 3 (4)
Dementia alzheimer's type (Nervous system disorders) | 0 (0) | 1 (1)
Demyelination (Nervous system disorders) | 1 (1) | 0 (0)
Diabetic autonomic neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Diabetic coma (Nervous system disorders) | 0 (0) | 1 (1)
Diabetic neuropathy (Nervous system disorders) | 6 (7) | 6 (6)
Dizziness (Nervous system disorders) | 6 (6) | 6 (6)
Dizziness postural (Nervous system disorders) | 0 (0) | 1 (1)
Embolic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 3 (3) | 4 (4)
Epilepsy (Nervous system disorders) | 4 (4) | 3 (3)
Essential tremor (Nervous system disorders) | 1 (1) | 0 (0)
Facial paralysis (Nervous system disorders) | 10 (10) | 6 (6)
Facial paresis (Nervous system disorders) | 1 (1) | 0 (0)
Generalised tonic-clonic seizure (Nervous system disorders) | 0 (0) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 2 (2) | 2 (2)
Haemorrhagic stroke (Nervous system disorders) | 4 (4) | 4 (4)
Haemorrhagic transformation stroke (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 1 (1)
Hemiparesis (Nervous system disorders) | 1 (1) | 3 (4)
Hepatic encephalopathy (Nervous system disorders) | 1 (2) | 0 (0)
Hypertensive encephalopathy (Nervous system disorders) | 3 (3) | 3 (3)
Hypoaesthesia (Nervous system disorders) | 2 (2) | 1 (1)
Hypotonia (Nervous system disorders) | 0 (0) | 1 (1)
Iiird nerve paralysis (Nervous system disorders) | 1 (1) | 1 (1)
Intracranial aneurysm (Nervous system disorders) | 0 (0) | 2 (2)
Intracranial mass (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic cerebral infarction (Nervous system disorders) | 0 (0) | 2 (2)
Ischaemic stroke (Nervous system disorders) | 30 (33) | 24 (24)
Lacunar infarction (Nervous system disorders) | 3 (3) | 7 (8)
Lacunar stroke (Nervous system disorders) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 3 (3) | 4 (4)
Lumbar radiculopathy (Nervous system disorders) | 3 (3) | 2 (2)
Lumbosacral plexus lesion (Nervous system disorders) | 1 (1) | 0 (0)
Lumbosacral radiculopathy (Nervous system disorders) | 1 (1) | 2 (2)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1)
Mental impairment (Nervous system disorders) | 1 (1) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 4 (4) | 1 (1)
Migraine (Nervous system disorders) | 2 (3) | 1 (1)
Monoplegia (Nervous system disorders) | 0 (0) | 1 (1)
Motor neurone disease (Nervous system disorders) | 2 (2) | 0 (0)
Multiple sclerosis (Nervous system disorders) | 2 (2) | 0 (0)
Multiple sclerosis relapse (Nervous system disorders) | 2 (4) | 0 (0)
Myasthenia gravis (Nervous system disorders) | 2 (6) | 0 (0)
Myelopathy (Nervous system disorders) | 1 (1) | 0 (0)
Myoclonus (Nervous system disorders) | 1 (1) | 0 (0)
Nerve compression (Nervous system disorders) | 0 (0) | 1 (1)
Nervous system disorder (Nervous system disorders) | 1 (1) | 1 (1)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (2)
Neurological symptom (Nervous system disorders) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 4 (4)
Normal pressure hydrocephalus (Nervous system disorders) | 0 (0) | 2 (2)
Paraesthesia (Nervous system disorders) | 0 (0) | 2 (2)
Paraparesis (Nervous system disorders) | 0 (0) | 1 (1)
Paraplegia (Nervous system disorders) | 1 (1) | 0 (0)
Parkinson's disease (Nervous system disorders) | 0 (0) | 2 (2)
Parkinsonism (Nervous system disorders) | 1 (1) | 1 (1)
Polyneuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 1 (1) | 1 (1)
Presyncope (Nervous system disorders) | 8 (8) | 5 (5)
Radial nerve palsy (Nervous system disorders) | 1 (1) | 0 (0)
Radicular pain (Nervous system disorders) | 1 (1) | 0 (0)
Radiculopathy (Nervous system disorders) | 6 (6) | 2 (2)
Sciatica (Nervous system disorders) | 4 (4) | 3 (3)
Seizure (Nervous system disorders) | 4 (4) | 5 (5)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Spinal cord compression (Nervous system disorders) | 0 (0) | 1 (1)
Spinal cord haematoma (Nervous system disorders) | 1 (1) | 0 (0)
Spinal cord herniation (Nervous system disorders) | 0 (0) | 1 (1)
Spinal cord infarction (Nervous system disorders) | 0 (0) | 1 (1)
Spinal cord ischaemia (Nervous system disorders) | 1 (1) | 0 (0)
Spinal vascular disorder (Nervous system disorders) | 0 (0) | 1 (1)
Spondylitic myelopathy (Nervous system disorders) | 1 (1) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 5 (5) | 3 (3)
Syncope (Nervous system disorders) | 32 (33) | 15 (16)
Thalamic infarction (Nervous system disorders) | 2 (2) | 1 (1)
Transient aphasia (Nervous system disorders) | 0 (0) | 1 (1)
Transient global amnesia (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 41 (46) | 41 (45)
Tremor (Nervous system disorders) | 1 (2) | 0 (0)
Vascular dementia (Nervous system disorders) | 3 (3) | 0 (0)
Vascular encephalopathy (Nervous system disorders) | 9 (9) | 1 (1)
Vascular headache (Nervous system disorders) | 1 (1) | 0 (0)
Vertebrobasilar insufficiency (Nervous system disorders) | 4 (4) | 2 (2)
Vertebrobasilar stroke (Nervous system disorders) | 0 (0) | 1 (1)
Vocal cord paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Device dislocation (Product Issues) | 1 (1) | 0 (0)
Device failure (Product Issues) | 0 (0) | 1 (1)
Device lead damage (Product Issues) | 0 (0) | 1 (1)
Device malfunction (Product Issues) | 0 (0) | 1 (1)
Device occlusion (Product Issues) | 2 (2) | 0 (0)
Device power source issue (Product Issues) | 1 (1) | 0 (0)
Thrombosis in device (Product Issues) | 0 (0) | 1 (1)
Acute psychosis (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (4) | 2 (2)
Anxiety disorder (Psychiatric disorders) | 0 (0) | 2 (3)
Bipolar disorder (Psychiatric disorders) | 0 (0) | 4 (5)
Borderline personality disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Completed suicide (Psychiatric disorders) | 2 (2) | 2 (2)
Confusional state (Psychiatric disorders) | 1 (1) | 2 (2)
Conversion disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 3 (3)
Depressed mood (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 10 (14) | 9 (11)
Depression suicidal (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Major depression (Psychiatric disorders) | 6 (7) | 3 (3)
Mania (Psychiatric disorders) | 0 (0) | 1 (1)
Mental disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 4 (4) | 5 (5)
Mood disorder due to a general medical condition (Psychiatric disorders) | 1 (1) | 0 (0)
Organic brain syndrome (Psychiatric disorders) | 0 (0) | 1 (1)
Post-traumatic stress disorder (Psychiatric disorders) | 1 (2) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Schizophrenia (Psychiatric disorders) | 1 (1) | 0 (0)
Stress (Psychiatric disorders) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 3 (4)
Acute kidney injury (Renal and urinary disorders) | 46 (54) | 53 (59)
Azotaemia (Renal and urinary disorders) | 0 (0) | 3 (3)
Bladder mass (Renal and urinary disorders) | 1 (1) | 0 (0)
Bladder outlet obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Bladder prolapse (Renal and urinary disorders) | 1 (1) | 0 (0)
Calculus bladder (Renal and urinary disorders) | 2 (2) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 3 (3) | 5 (5)
Chronic kidney disease (Renal and urinary disorders) | 15 (16) | 7 (8)
Cystitis haemorrhagic (Renal and urinary disorders) | 0 (0) | 1 (1)
Diabetic nephropathy (Renal and urinary disorders) | 3 (3) | 2 (2)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
End stage renal disease (Renal and urinary disorders) | 4 (6) | 9 (10)
Genitourinary symptom (Renal and urinary disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 8 (8) | 6 (9)
Hydronephrosis (Renal and urinary disorders) | 6 (6) | 2 (2)
Hypertensive nephropathy (Renal and urinary disorders) | 1 (1) | 0 (0)
Hypertonic bladder (Renal and urinary disorders) | 1 (1) | 0 (0)
Ketonuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Lower urinary tract symptoms (Renal and urinary disorders) | 0 (0) | 2 (2)
Nephrolithiasis (Renal and urinary disorders) | 15 (18) | 20 (24)
Nephropathy (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrotic syndrome (Renal and urinary disorders) | 2 (2) | 1 (1)
Renal artery arteriosclerosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal artery stenosis (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal artery thrombosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal colic (Renal and urinary disorders) | 3 (4) | 3 (3)
Renal cyst (Renal and urinary disorders) | 1 (1) | 2 (2)
Renal embolism (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 17 (18) | 16 (17)
Renal haematoma (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal haemorrhage (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 6 (6) | 2 (2)
Renal injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal ischaemia (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal mass (Renal and urinary disorders) | 2 (2) | 1 (1)
Stag horn calculus (Renal and urinary disorders) | 0 (0) | 1 (1)
Stress urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 (1) | 0 (0)
Ureteric stenosis (Renal and urinary disorders) | 2 (2) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 8 (9) | 8 (9)
Urethral haemorrhage (Renal and urinary disorders) | 0 (0) | 1 (1)
Urethral stenosis (Renal and urinary disorders) | 2 (2) | 0 (0)
Urinary bladder haemorrhage (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary fistula (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 2 (2)
Urinary retention (Renal and urinary disorders) | 6 (7) | 5 (5)
Acquired hydrocele (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Adenomyosis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Adnexal torsion (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Balanoposthitis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 11 (13) | 18 (18)
Breast discharge (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Breast disorder (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Breast hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Breast mass (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Endometrial hyperplasia (Reproductive system and breast disorders) | 4 (4) | 0 (0)
Endometrial thickening (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Endometriosis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Epididymal cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Female genital tract fistula (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Genital leukoplakia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Haemorrhagic ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Pelvic congestion (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pelvic fluid collection (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pelvic prolapse (Reproductive system and breast disorders) | 3 (3) | 0 (0)
Perineal cyst (Reproductive system and breast disorders) | 1 (2) | 0 (0)
Peyronie's disease (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 4 (4) | 1 (1)
Prostatic disorder (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Prostatomegaly (Reproductive system and breast disorders) | 0 (0) | 2 (3)
Seminal vesiculitis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Spermatocele (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Testicular cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Testicular mass (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Uterine polyp (Reproductive system and breast disorders) | 1 (1) | 2 (2)
Uterine prolapse (Reproductive system and breast disorders) | 2 (2) | 3 (3)
Vaginal fistula (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal prolapse (Reproductive system and breast disorders) | 2 (2) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 23 (29) | 15 (16)
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 11 (11)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 31 (35) | 38 (42)
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 15 (17)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Epiglottic cyst (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 13 (13) | 7 (7)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypersensitivity pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pharyngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pickwickian syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 6 (8) | 7 (7)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 23 (23) | 20 (20)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (5)
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 4 (6)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 12 (17)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 7 (7)
Tonsillar disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Vocal cord polyp (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acanthosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Alopecia scarring (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Dermatomyositis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 6 (7) | 14 (16)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Granuloma annulare (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Henoch-schonlein purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hidradenitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypersensitivity vasculitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Ischaemic skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Panniculitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin necrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 8 (9) | 12 (14)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Aborted pregnancy (Social circumstances) | 1 (1) | 0 (0)
Hospitalisation (Surgical and medical procedures) | 1 (1) | 0 (0)
Accelerated hypertension (Vascular disorders) | 1 (1) | 1 (1)
Aneurysm (Vascular disorders) | 0 (0) | 2 (2)
Aortic aneurysm (Vascular disorders) | 16 (16) | 11 (12)
Aortic aneurysm rupture (Vascular disorders) | 2 (2) | 0 (0)
Aortic dissection (Vascular disorders) | 5 (5) | 2 (2)
Aortic embolus (Vascular disorders) | 1 (1) | 0 (0)
Aortic stenosis (Vascular disorders) | 8 (8) | 4 (5)
Arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0)
Arterial stenosis (Vascular disorders) | 1 (1) | 0 (0)
Arteriosclerosis (Vascular disorders) | 3 (3) | 2 (2)
Blood pressure inadequately controlled (Vascular disorders) | 0 (0) | 1 (1)
Circulatory collapse (Vascular disorders) | 3 (3) | 3 (4)
Deep vein thrombosis (Vascular disorders) | 14 (15) | 15 (16)
Diabetic vascular disorder (Vascular disorders) | 2 (3) | 1 (1)
Dry gangrene (Vascular disorders) | 0 (0) | 2 (2)
Embolism (Vascular disorders) | 0 (0) | 1 (1)
Embolism venous (Vascular disorders) | 1 (1) | 1 (1)
Essential hypertension (Vascular disorders) | 1 (1) | 1 (2)
Extremity necrosis (Vascular disorders) | 2 (2) | 5 (6)
Femoral artery perforation (Vascular disorders) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 5 (5) | 0 (0)
Haemodynamic instability (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 30 (33) | 31 (35)
Hypertensive crisis (Vascular disorders) | 15 (19) | 9 (12)
Hypertensive emergency (Vascular disorders) | 1 (1) | 4 (4)
Hypertensive urgency (Vascular disorders) | 6 (6) | 4 (4)
Hypotension (Vascular disorders) | 11 (11) | 10 (12)
Hypovolaemic shock (Vascular disorders) | 1 (1) | 4 (4)
Iliac artery occlusion (Vascular disorders) | 0 (0) | 3 (3)
Iliac artery stenosis (Vascular disorders) | 3 (3) | 2 (2)
Inferior vena cava perforation (Vascular disorders) | 1 (1) | 0 (0)
Intermittent claudication (Vascular disorders) | 4 (4) | 4 (7)
Jugular vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Leriche syndrome (Vascular disorders) | 1 (1) | 0 (0)
Lymphoedema (Vascular disorders) | 2 (2) | 3 (3)
Malignant hypertension (Vascular disorders) | 0 (0) | 1 (1)
Neurogenic shock (Vascular disorders) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 4 (4) | 10 (11)
Peripheral arterial occlusive disease (Vascular disorders) | 30 (39) | 45 (52)
Peripheral artery aneurysm (Vascular disorders) | 3 (4) | 3 (4)
Peripheral artery aneurysm rupture (Vascular disorders) | 1 (1) | 0 (0)
Peripheral artery occlusion (Vascular disorders) | 7 (8) | 8 (10)
Peripheral artery stenosis (Vascular disorders) | 7 (8) | 3 (5)
Peripheral artery thrombosis (Vascular disorders) | 4 (4) | 1 (2)
Peripheral coldness (Vascular disorders) | 1 (1) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 16 (21) | 11 (13)
Peripheral vascular disorder (Vascular disorders) | 13 (20) | 12 (16)
Peripheral venous disease (Vascular disorders) | 0 (0) | 1 (1)
Phlebitis (Vascular disorders) | 1 (1) | 1 (1)
Shock (Vascular disorders) | 0 (0) | 1 (1)
Subclavian artery stenosis (Vascular disorders) | 1 (1) | 0 (0)
Subclavian steal syndrome (Vascular disorders) | 1 (1) | 0 (0)
Subclavian vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Thrombophlebitis (Vascular disorders) | 1 (1) | 3 (3)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Vasculitis (Vascular disorders) | 1 (1) | 1 (1)
Venous thrombosis limb (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Epanova (N=6532) | Placebo (N=6535)
Abdominal discomfort (Gastrointestinal disorders) | 87 (102) | 35 (38)
Abdominal pain (Gastrointestinal disorders) | 90 (104) | 54 (61)
Abdominal pain upper (Gastrointestinal disorders) | 80 (99) | 59 (68)
Diarrhoea (Gastrointestinal disorders) | 765 (1049) | 316 (386)
Dyspepsia (Gastrointestinal disorders) | 89 (104) | 41 (53)
Nausea (Gastrointestinal disorders) | 204 (229) | 110 (126)
Nasopharyngitis (Infections and infestations) | 97 (193) | 75 (145)
Diabetes mellitus (Metabolism and nutrition disorders) | 147 (150) | 121 (122)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 130 (131) | 153 (155)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Principal Investigator shall provide AstraZeneca with copies of any materials relating to the Study, the Study Documentation, or the Developed Technologies that either Party intends to publish (or submit for publication) or make any presentations relating to, at least 60 days in advance of publication, submission or presentation.

DOCUMENTS (2):
  • Study Protocol (2015-05-01): https://cdn.clinicaltrials.gov/large-docs/17/NCT02104817/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-22): https://cdn.clinicaltrials.gov/large-docs/17/NCT02104817/SAP_001.pdf